CLINICAL TRIAL: NCT01360840
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Trial Investigating Two Doses of EMD 525797 in Subjects With Asymptomatic or Mildly Symptomatic Metastatic Castrate-resistant Prostate Cancer (mCRPC)
Brief Title: EMD 525797 in Subjects With Asymptomatic or Mildly Symptomatic Metastatic Castrate-resistant Prostate Cancer
Acronym: PERSEUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 62242-006
Record Dates: First submitted 2011-04-15; First posted 2011-05-26 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer Metastatic
Keywords: Asymptomatic; mildly symptomatic; metastatic castrate-resistant prostate cancer; mCRPC
MeSH Terms: interventions — Abituzumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + Standard of care (SoC) (Placebo Comparator)
  Interventions: Other: Placebo; Other: Standard of Care (SoC)
- EMD 525797 750 mg + SoC (Experimental)
  Interventions: Drug: EMD 525797; Other: Standard of Care (SoC)
- EMD 525797 1500 mg + SoC (Experimental)
  Interventions: Drug: EMD 525797; Other: Standard of Care (SoC)

INTERVENTIONS:
Drug: EMD 525797 — Subjects will be administered with EMD 525797 at a dose of 1500 milligram (mg) (diluted with 0.9 percent [%] sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons.
  Arms: EMD 525797 1500 mg + SoC
Drug: EMD 525797 — Subjects will be administered with EMD 525797 at a dose of 750 mg (diluted with 0.9% sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons.
  Arms: EMD 525797 750 mg + SoC
Other: Placebo — Subjects will be administered with placebo (as 0.9% sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons.
  Arms: Placebo + Standard of care (SoC)
Other: Standard of Care (SoC) — All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists).

SUMMARY:
The primary objective of the trial is to evaluate the clinical anti-tumor activity of EMD 525797 administered as 1-hour intravenous infusion every 3 weeks in terms of progression free survival (PFS) time in subjects with asymptomatic or mildly symptomatic metastatic castrate-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate (Gleason score)
* Bisphosphonate treatment
* Stable, ongoing adequate testosterone suppression proven by hypogonadal levels of testosterone (less than or equal to) <= 50 nanogram per deciliter [ng/dL]) for subjects without surgical castration (luteinizing hormone-releasing hormone antagonists and agonists)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior chemotherapy, biologic therapy (targeted therapy), or any experimental therapy for mCRPC
* Chronic and ongoing treatment with opioids
* Acute pathologic fracture, spinal cord compression, or hypercalcemia at Screening
* Visceral metastasis, brain metastasis
* Radiotherapy to bone lesions and/or orthopedic surgery for pathologic fractures. Any kinds of major elective surgery within 30 days prior to trial treatment
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (71):
- United States (12):
  - Research Site, Pleasant Hill, California
  - Research Site, Chicago, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, Cleveland, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Roanoke, Virginia
  - Research Site, Spokane, Washington
- Australia (10):
  - Research Site, Bendigo
  - Research Site, Coffs Harbour
  - Research Site, Darlinghurst
  - Research Site, Frankston
  - Research Site, Gosford
  - Research Site, Kurralta Park
  - Research Site, Northmead
  - Research Site, Port Macquarie
  - Research Site, Randwick
  - Research Site, Turnhout
- ZNA Middelheim Oncologie, Antwerp, Belgium
- Canada (6):
  - Brandord Urology Research, Brantford, Ontario
  - Exdeo Clinical Research Inc., Abbotsford
  - Can-Med Clinical Research Inc., Province of British Columbia
  - Sunnybrook Health Sciences Centre, Toronto
  - Research Site, Victoria
  - Research Site, Windsor
- France (7):
  - Research Site, Angers
  - Center Alexis Vaurrin, Bourgogne
  - Research Site, Caen
  - Hôpitaux Civils de Colmar-CH Louis Pasteur, Colmar
  - Research Site, Paris
  - Research Site, Reims
  - Institute Gustave Roussy, Villejuif
- Germany (10):
  - Research Site, Aachen
  - Universitätsmedizin Charité, Campus Benjamin Franklin, Urologische Klinik and Poliklinik, Berlin
  - Research Site, Darmstadt
  - Universitätsklinikum Carl Gustav Carus an der Techischen Universität Dresden, Klinik und Poliklinik für Urologie, Dresden
  - Research Site, Esslingen am Neckar
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, Nürtingen
  - Studienpraxis Urologie, Reutlingen
  - Universitätsklinikum Tübinger, Klinik und Poliklinik für Urologie, Tübingen
- Netherlands (3):
  - Research Site, Blaricum
  - Research Site, Groningen
  - Research Site, Haarlem
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Lublin
- Russia (10):
  - Altay Regional Oncology Dispensary, Barnaul
  - Research Site, Barnaul
  - State Institution of Healthcare Ivanovo Regional Oncology Dispensary, Ivanovo
  - Budzhet Clinical Oncology Center, Izhevsk
  - Research Site, Kazan'
  - Krasnoyarsk State Medical University Oncology and Radiotherapy Territorial Dispensary, Krasnoyarsk
  - Research Site, Omsk
  - City Hospital # 2, Saint Petersburg
  - Research Site, Stavropol
  - Research Site, Yekaterinburg
- Research Site, Prešov, Slovakia
- South Africa (4):
  - Research Site, Gauteng
  - Research Site, Kwa-Zulu Natal
  - Research Site, Pretoria Gauteng
  - Research Site, Western Cape
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Sabadell, Barcelone

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): April 2011/December 2012. Study completion date: July 2014. Clinical data cut-off: 30 April 2013. Subjects were recruited in 11 countries (Australia, Belgium, Canada, France, Germany, Netherlands, Poland, Russia, South Africa, Spain, and USA) across the globe in 65 centers.
Pre-assignment Details: Enrolled: 283 screened for eligibility; 103 were excluded (mainly non-fulfillment of inclusion or exclusion criteria). 180 subjects were assigned to the treatment groups. Two subjects did not receive study drug administration.
Groups:
- Placebo + SoC: Subjects were administered with placebo 0.9% sodium chloride as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the standard of care (SoC) consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
- EMD 525797 750 mg + SoC: Subjects were administered with EMD 525797 at a dose of 750 mg (diluted with 0.9% sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
- EMD 525797 1500 mg + SoC: Subjects were administered with EMD 525797 at a dose of 1500 mg (diluted with 0.9% sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
Period: Overall Study
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Started | 60 | 60 | 60
Completed | 50 | 50 | 51
Not Completed | 10 | 10 | 9
Not completed — Ongoing at data cut-off | 10 | 10 | 9

BASELINE CHARACTERISTICS:
Population: All Subjects (ALL) analysis set included subjects who signed the Informed consent document.
Groups:
- Placebo + SoC: Subjects were administered with placebo 0.9% sodium chloride as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
- Total: Total of all reporting groups
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.43) | 69.0 (7.31) | 70.0 (8.88) | 69.6 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Time
Description: PFS was defined as time from randomization until the first documented sign of objective radiographic disease progression (ORDP) or death from any cause. Death was considered as an event only if it was reported within 12 weeks after last tumor assessment without progression. ORDP was defined as: Bone lesion progression (2 or more new bone lesions compared to baseline) assessed with bone scintigraphy. Assessment was based on Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) modified as per Prostate Cancer Working Group 2 (PCWG-2); Soft-tissue lesion progression assessed with CT scans according to RECIST v1.0 modified as per PCWG-2; Presence of skeletal events defined as cord compression/fracture documented via a scheduled or unscheduled radiographic assessment triggered by increased pain or other signs and/or symptoms, based on the investigator's discretion; Non-radiological events, including emergency bone irradiation and surgery, were not investigated.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: Intention-to-treat (ITT) analysis set included all the subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
months | 3.3 [2.8 to 4.8] | 3.4 [2.8 to 5.6] | 4.3 [2.8 to 6.6]
Statistical Analysis 1: Comparison: Placebo + SoC vs EMD 525797 750 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.57 to 1.39]
Statistical Analysis 2: Comparison: Placebo + SoC vs EMD 525797 1500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.52 to 1.26]

2. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
months | NA [14.8 to NA] — The value was not estimable due to lack of events | NA [12.9 to NA] — The value was not estimable due to lack of events | NA [14.4 to NA] — The value was not estimable due to lack of events
Statistical Analysis 1: Comparison: Placebo + SoC vs EMD 525797 750 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.52 to 2.31]
Statistical Analysis 2: Comparison: Placebo + SoC vs EMD 525797 1500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.47 to 2.15]

3. Secondary Outcome: Time to Tumor Progression
Description: Time to tumor progression was defined as the time from the date of randomization to the date of ORDP. ORDP was defined as: Bone lesion progression (2 or more new bone lesions compared to baseline) assessed with bone scintigraphy, which had to be confirmed by bone scintigraphy 6 weeks later if subjects remained asymptomatic or mildly symptomatic. Assessments were to be based on RECIST v1.0 modified according to PCWG-2; Soft-tissue lesion progression assessed with CT scans according to RECIST v1.0 modified as per PCWG-2; Presence of skeletal events defined as cord compression or fracture documented via a scheduled or unscheduled radiographic assessment triggered by increased pain or other signs and/or symptoms, based on the investigator's discretion; Non-radiological events, including emergency bone irradiation and surgery, were not investigated.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
months | 3.3 [2.8 to 5.4] | 3.4 [2.8 to 5.6] | 4.6 [2.8 to 6.9]
Statistical Analysis 1: Comparison: Placebo + SoC vs EMD 525797 750 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.58 to 1.44]
Statistical Analysis 2: Comparison: Placebo + SoC vs EMD 525797 1500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.52 to 1.27]

4. Secondary Outcome: Number of Subjects With Presence of Tumor Response and Disease Control (DC) in Soft Tissue Lesions
Description: Presence of tumor response in soft tissue lesions was defined as the presence of at least 1 confirmed complete response (CR) or confirmed partial response (PR) in soft tissue lesions, documented by computed tomography (CT) scans. Presence of DC in soft tissue lesions was defined as the presence of at least 1 confirmed CR or confirmed PR or stable disease (SD) lasting at least 12 weeks after randomization. Tumor response assessments were based on RECIST v1.0 modified according to the PCWG-2. The response was evaluated for subjects with measurable disease at baseline. According to RECIST v1.0, CR=disappearance of all target and non-target lesions; PR=at least 30% decrease in the sum of the longest diameter of target lesions and non-complete response/non-progressive disease in non-target lesions.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects who were randomized in the study. "N" signifies the total number of subjects evaluable for this outcome measure.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 28 | 22 | 24
Subjects
  Tumor response | 1 | 0 | 1
  Disease control | 2 | 3 | 4

5. Secondary Outcome: Number of Subjects With New Bone Lesions Compared to Baseline
Description: New bone lesions were evaluated by bone scintigraphy for subjects with bone lesions at baseline.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects randomized in the study. "N" signifies the total number of subjects evaluable for this outcome measure.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 57 | 57 | 57
Subjects | 40 | 34 | 34

6. Secondary Outcome: Number of Subjects With Presence of DC in Bone Lesions
Description: Presence of DC in bone lesions was defined as the appearance of less than 2 new bone lesions, documented by bone scintigraphy.
Time Frame: At Weeks 13, 19 and 25
Population: ITT analysis set included all the subjects randomized in the study.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
Subjects
  Week 13 | 4 | 7 | 7
  Week 19 | 2 | 7 | 6
  Week 25 | 2 | 4 | 3

7. Secondary Outcome: Bone and Soft Tissue Lesions Composite Tumor Response
Description: Bone and soft tissue lesions composite tumor response was defined as the presence of both a confirmed CR or PR, documented by CT scans, and a DC in bone lesions, documented by bone scintigraphy. CR was defined as disappearance of all target and non-target lesions and PR was defined as at least 30% decrease in the sum of the longest diameter of target lesions and non-complete response/non-progressive disease in non-target lesions. Presence of DC in bone lesions was defined as the appearance of less than 2 new bone lesions.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects who were randomized in the study.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
Subjects | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects With Presence of Skeletal Related Events
Description: Presence of skeletal related events was defined as cord compression or fracture documented via a scheduled or unscheduled radiographic assessment triggered by increased pain or other signs and/or symptoms at the investigator discretion. Non-radiological events, including emergency bone irradiation and surgery, were not investigated.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: ITT analysis set included all the subjects who were randomized in the study.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 60 | 60
Subjects | 2 | 8 | 3

9. Secondary Outcome: Number of Subjects With Presence of Prostate Specific Antigen (PSA) Response
Description: PSA response was defined as a decrease greater than 50 percent (%) in PSA value from baseline for 2 consecutive evaluations greater than or equal to (>=) 3 Weeks apart.
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 58 | 60
Subjects | 3 | 6 | 5

10. Secondary Outcome: Minimum Percentage Change From Baseline in PSA Serum Concentration
Time Frame: Baseline, up to data cut-off date (30 April 2013), assessed up to 2 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 58 | 57 | 60
Percent change | 24.00 (86.156) | 35.65 (127.677) | 14.70 (50.841)

11. Secondary Outcome: Minimum Percentage Change From Baseline in the Number of Circulating Tumor Cells (CTCs)
Time Frame: Time from randomization until data cut-off date (30 April 2013), assessed up to 2 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 29 | 27 | 22
Percent change | 49.02 (127.643) | 354.74 (1038.195) | 280.58 (482.653)

12. Secondary Outcome: Overall Minimum Percentage Change From Previous Time Point in Circulating Tumor Cells (CTC)
Time Frame: Cycle 1, Day 1 (Week 1): pre-dose, Cycle 3, Day 1 (Week 7): pre-dose, and Cycle 5, Day 1 (Week 13): pre-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 36 | 34 | 30
Percent change | 9.54 (103.225) | 223.97 (868.941) | 179.11 (446.428)

13. Secondary Outcome: Number of Subjects With Any Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, and TEAEs Leading to Discontinuation
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were defined as those AEs that started between first dose of study drug and up to 50 days after last dose.
Time Frame: From the first dose of study drug administration until 50 days after the last dose of study drug administration or until cut-off date (30 April 2013), assessed up to 2 years
Population: The Safety analysis set included all the randomized subjects who received at least 1 dose of planned trial treatment and had at least one safety assessment following the trial treatment.
Measure: Number; unit: Subjects
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 60 | 58 | 60
Subjects
  TEAEs | 55 | 49 | 53
  Serious TEAEs | 16 | 13 | 14
  TEAEs leading to death | 2 | 2 | 3
  TEAEs Leading to Permanent Discontinuation | 5 | 11 | 8

14. Secondary Outcome: Pharmacokinetic Parameter: Clearance of Intravenously Administered EMD 525797 After First Dose (CL) and Clearance in Steady State of EMD52597 After Fifth Dose (CLss)
Description: The apparent total body clearance of drug following intravenous administration (CL); The apparent total body clearance of drug at steady state following intravenous administration (CLss).
Time Frame: Cycle 1 (Week 1) and cycle 5 (Week 13): Day 1: pre-dose, End of Infusion (EOI), 4, 8, 24, 48, 96, 168, 336, and 504 hours after start of infusion; Cycles 3 and 4 (Weeks 7 and 10), Day 1: pre-dose; Cycle 7 (Week 19), Day 1: pre-dose and EOI
Population: Pharmacokinetic Analysis Set (PKA) included all the randomized subjects who received at least the first dose of the trial drug and provided sufficient data for a concentration time profile for EMD 525797. "n" signifies the number of subjects evaluable for each category in the evaluated group, respectively.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 4 | 6
Liter per hour
  First dose: CL (n=4, 6) | 0.017 (0.007) | 0.013 (0.003)
  Fifth dose: CLss (n=2, 4) | 0.017 (0.002) | 0.010 (0.001)

15. Secondary Outcome: Pharmacokinetic Parameter: Volume of Distribution of EMD 525797 After the First Dose (V) and in Steady State After the Fifth Dose (Vss) of Intravenous Infusion
Description: The apparent volume of distribution during the terminal phase following intravenous administration (V). The estimate of the apparent volume of distribution at steady state following intravenous administration (Vss).
Time Frame: as for outcome 14
Population: PKA included all the randomized subjects who received at least the first dose of the trial drug and provided sufficient data for a concentration time profile for EMD 525797. "n" signifies the number of subjects evaluable for each category in the evaluated group, respectively.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 4 | 6
liter
  First dose (n=4, 6) | 4.55 (1.02) | 4.60 (0.74)
  Fifth dose (n=2, 4) | 4.81 (NA) — The sample size of n=2 was inappropriate for Vss parameter to calculate standard deviation. Hence, it was not calculated. | 5.18 (0.56)

16. Other Pre Specified Outcome: To Explore the Relationship Between Number and/or Changes of Numbers of Biomarker and the Clinical Outcome
Time Frame: From the date of randomization up to data cut-off date (30 April 2013), assessed up to 2 years
Population: Data for this outcome measure was presented graphically as per planned analysis but not statistically summarized.
Arm/Group | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration until 50 days after the last dose of study drug administration or until cut-off date (30 April 2013), assessed up to 2 years
Groups:
- Placebo + SoC: Subjects were administered with placebo 0.9 percent (%) sodium chloride as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
- EMD 525797 750 mg + SoC: Subjects were administered with EMD 525797 at a dose of 750 milligram (mg) (diluted with 0.9% sodium chloride) as a 1-hour intravenous infusion every 3 Weeks until disease progression or unacceptable toxicity, whichever comes first, unless the subject stopped the trial treatment for other reasons. All the subjects followed the SoC consisting of the continued treatment with luteinizing-hormone releasing hormone agonists (or antagonists). In order to avoid any confounding effects, bisphosphonate treatment was initiated 2 days before start of treatment with EMD 525797.
Arm/Group | Placebo + SoC | EMD 525797 750 mg + SoC | EMD 525797 1500 mg + SoC
Serious Adverse Events (participants affected / at risk) | 16/60 | 13/58 | 14/60
Other Adverse Events (participants affected / at risk) | 53/60 | 47/58 | 53/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + SoC (N=60) | EMD 525797 750 mg + SoC (N=58) | EMD 525797 1500 mg + SoC (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Epiduritis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Orthostatis hypotension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + SoC (N=60) | EMD 525797 750 mg + SoC (N=58) | EMD 525797 1500 mg + SoC (N=60)
Anaemia (Blood and lymphatic system disorders) | 10 | 6 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2
Eye pain (Eye disorders) | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Asthenopia (Eye disorders) | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 3
Nausea (Gastrointestinal disorders) | 2 | 6 | 6
Constipation (Gastrointestinal disorders) | 7 | 6 | 3
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1
Periodonditis (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
oral pain (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 12 | 10 | 9
Influenza like illness (General disorders) | 4 | 8 | 3
Asthenia (General disorders) | 9 | 3 | 6
oedema peripheral (General disorders) | 1 | 7 | 1
Pyrexia (General disorders) | 2 | 4 | 4
Pain (General disorders) | 1 | 2 | 3
Chest pain (General disorders) | 0 | 2 | 1
Spinal pain (General disorders) | 1 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Crying (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 3 | 1 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 2
Anal fungal infection (Infections and infestations) | 0 | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 4 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Perineal infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Weight decreased (Investigations) | 6 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 4
Blood creatinine increased (Investigations) | 1 | 2 | 3
Fibrin D dimer increased (Investigations) | 4 | 2 | 3
C-reactive protein increased (Investigations) | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Blood potassium increased (Investigations) | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 0
Calcium ionised decreased (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 1 | 0
Gamma-glutamyl transferase increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 8 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumor invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 5 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1 | 0
Cervical root pain (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Epiduritis (Nervous system disorders) | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Paresis (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 3
Depression (Psychiatric disorders) | 1 | 1 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 4 | 3
Proteinuria (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Renal and urinary disorders) | 0 | 1 | 1
Balanitis (Renal and urinary disorders) | 0 | 1 | 0
Penile pain (Renal and urinary disorders) | 0 | 1 | 0
Perineal pain (Renal and urinary disorders) | 0 | 0 | 1
Gynaecomastia (Renal and urinary disorders) | 1 | 0 | 0
Testicular pain (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 3 | 2 | 2
Hypertension (Vascular disorders) | 3 | 1 | 2
Hypotension (Vascular disorders) | 2 | 2 | 1
Orthostatic hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other